CLINICAL TRIAL: NCT01862341
Title: The Effect of Milk Powder With Fiber and Probiotics on Digestive Habits and General Health Well-being of Selected Filipino Mothers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fonterra Research Centre (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FON-JOLIE-PPH-2012-01
Record Dates: First submitted 2013-05-10; First posted 2013-05-24 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Constipation
Keywords: Constipation; Bowel movement; Intestinal health
MeSH Terms: conditions — Constipation

ARMS (1):
- Milk powder (Experimental): ANMUM In-Shape Nutritional Milk Powder for Active Mothers. The dose of the milk powder is 40g added to 200ml of drinkable water and will be taken twice a day.
  Interventions: Dietary Supplement: ANMUM In-Shape Nutritional Milk Powder for Active Mothers

INTERVENTIONS:
Dietary Supplement: ANMUM In-Shape Nutritional Milk Powder for Active Mothers

SUMMARY:
In-Shape Nutritional Milk Powder is a nutritional milk powder containing fibers, probiotics and other nutrients. This study will focus on the effects of fiber and probiotics on digestive health and health well being in selected Filipino mothers

ELIGIBILITY:
Inclusion Criteria:

* Female between 21 and 35 years of age.
* Has at least one child under the age of three.
* Willingness and ability to participate in the study.
* Suffering from mild to moderate constipation and bowel troubles, and non-specific symptoms including bloating, flatulence, gurgling, feeling heavy after eating, and abdominal pain.
* Slow transit or irregular bowels movements (stool consistency harder than usual or fewer bowel movements, i.e. every 2-3 days or less than 3 bowel movements per week).
* Agree to maintain dietetic measures (on their own volition or as previously recommended by health/nutrition professionals), if any, during the study period.
* Subject, or subject's legally acceptable representative, has voluntarily signed and dated an informed consent form, approved by a local Ethics Committee/Institutional Review Board authorization prior to any participation in the study.

Exclusion Criteria:

* Having participated in another trial currently and up to two months prior to this trial date.
* Known chronic constipation.
* Treated gastrointestinal symptoms.
* Regular intake of laxatives or other remedies to promote digestion (herbal teas, peppermint etc.) during the two weeks before the start of the study or during the study.
* Consuming dairy products or supplements containing Probiotics (e.g., yogurt, Lactic acid drink, drinkable yogurt, food supplements, extracts), Prebiotics (e.g., Oligosaccharides), or fiber supplements within 10 days prior to the start of the study or during the study.
* Currently taking (and during the past 3 months) any dietary fiber supplementation except from food sources.
* Previous contraindication to fiber supplement (Crohn's disease).
* Recently or currently on antibiotic medication in the past two weeks.
* Known allergy to milk proteins or intolerance to lactose.
* Currently pregnant.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Bowel improvement | up to day 28
  Evaluate the perceptions of selected Filipino women (21-35 years of age) on the effectiveness of milk powder with fiber and probiotics on improving bowel movement through questionnaires.

SECONDARY OUTCOMES:
Intestinal health | Day 0 and day 28
  Assess intestinal improvement determined by questionnaire on sensation after bowel movement and state of stools (color, odor, shape) through a questionnaire.
General well-being and lifestyle attitudes | Day 3, 7, 10, 14, 21, 24, and 28
  Assess the general well-being and lifestyle attitudes through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Imelda Agdeppa, PhD, Principal Investigator — FNRI
Locations (4):
- Philippines (4):
  - Camp Bagong Diwa, City of Taguig
  - Villamor Air Base, Makati
  - Camp Aguinaldo, Manila
  - Camp Crame, Quezon